CLINICAL TRIAL: NCT05135299
Title: Complications in Acute Calculous Cholecystitis
Status: Completed | Type: Observational
Sponsor: Hospital del Mar (Other)
Responsible Party: Principal Investigator, Ana María González Castillo, Principal Investigator, Hospital del Mar
Other Study IDs: Complications in ACC
Record Dates: First submitted 2021-05-14; First posted 2021-11-26 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Acute Calculous Cholecystitis
Keywords: Emergent Cholecystectomy; Mortality in acute cholecystitis; High Risk Patient; Morbidity in Acute Cholecystitis; Risk Factors in Acute Cholecystitis; Unfit for Surgery; Acute Cholecystitis; Acute Calculous Cholecystitis
MeSH Terms: conditions — Cholecystitis, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute calculous cholecystitis (ACC) is the second most frequent surgical condition in emergency departments, the complication rate of ACC is 8-20%, and the mortality rate is 0.5-6% in recent series. The Tokyo Guidelines (TG) advocate for different risk factors and initial treatments of ACC with no clear evidence that all patients will benefit from them.

The objective of the study is to identify the risk factors for complications in ACC.

It is a retrospective cohort study conducted from January 2011 to December 2016 in a single center with a dedicated surgical emergency unit in a Metropolitan University Hospital in Barcelona, Spain. The analysis of the data was finished in March 2020.

The study candidates comprised 963 consecutive patients with a diagnosis of ACC according to the TG18 and/or received a diagnosis of ACC in the Pathology report in those that an emergent cholecystectomy was performed.

The study case definition was a 'Pure Acute Cholecystitis' (pure ACC); therefore, patients with any other concomitant diagnosis potentially influencing outcome (Postoperative cholecystitis, Acute Cholangitis, Acute Pancreatitis, Incidental Cholecystectomy, Acalculous Cholecystitis, Chronic Cholecystitis/Persistent Colic, Post-endoscopic retrograde pancreato-cholangiography, or Neoplasia) were excluded from the final analysis.

Variables:

Primary data were available from a prospective database maintained in File Maker v.12 (Mountainview, CA, USA), which included basic demographic data, type of interventions, sex, days of admission, and complications. Every record was completed by browsing the electronic patient record, adding laboratory and microbiology data, as well as antibiotic therapy, duration of procedure, additional procedures, and grade of acute cholecystitis according to the TG18 diagnostic criteria.

Preoperative comorbidities were assessed using the Charlson Comorbidity Index and surgical risk by ASA classification. The type of initial treatment was classified as Surgical Treatment (Cholecystectomy either by laparoscopy or laparotomy) or Non-Surgical Treatment, which was either percutaneous cholecystostomy or intravenous antibiotics alone.

The main outcome measure was the mortality after the diagnostic of ACC. In the patients that were discharged, 30 days after the diagnosis, if the patients was not discharged in 30 days, at any time during the same admission.

Interventions:

All patients received intravenous antibiotic therapy from the moment the diagnosis was formulated, according to a fixed protocol.

Ultrasound-guided cholecystostomy was performed percutaneously with an 8-Fr catheter (SKATER ™, Argon Medical Devices, Rochester, NY, USA) by either transhepatic or transperitoneal insertion, at the discretion of the radiologist.

Laparoscopic Cholecystectomy was performed according to the French technique using 4 trochars. The content of the gallbladder was evacuated by Veress needle puncture when necessary.

Statistical Analysis:

The discrimination power of the model was assessed by receiver operating characteristic (ROC) curves and was compared with the DeLong method.

Legal and Ethical considerations This study was approved by the clinical research ethical committee of the Hospital del Mar and was classified as a non-clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic of a "Pure" Acute Calculous Cholecystitis.
* Older than 18 years old.

Exclusion Criteria:

* Younger than 18 years old.
* Any concomitant diagnostic that could change the prognostic of a "Pure" ACC, for example: Cholangitis, Pancreatitis, Postoperative ACC, Acalculous cholecystitis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients admited with a diagnostic of Acute Cholecystitis in a dedicated surgical emergency unit, from January 2011 to December 2016, in a Metropolitan University Hospital in Barcelona, Spain.
Sampling Method: Probability Sample
Enrollment: 963 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2021-04 (Actual)

PRIMARY OUTCOMES:
Number of patients withs complications after diagnosis of Acute Calculous Cholecystitis | 2011-2016
  The main outcome measure was the total of complications in patients with an Acute Calculous Cholecystitis assessed by the Clavien-Dindo Classification.
Description of the risk factors for complications with the demographic data | 2011-2016
  We will study the increased risk of an event associated with a variable reported as the Odds Ratio (OR) and 95% confidence interval (CI) of the gender (Male/Female)
Description of the risk factors for complications with the demographic data | 2011-2016
  We will study the increased risk of an event associated with a variable reported as the Odds Ratio (OR) and 95% confidence interval (CI) of the age in years.
Description of the risk factors for complications with the physiological parameters | 2011-2016
  We will study the increased risk of an event associated with a variable reported as the Odds Ratio (OR) and 95% confidence interval (CI) of the temperature in Celsius.
Description of the risk factors for complications with the physiological parameters | 2011-2016
  We will study the increased risk of an event associated with a variable reported as the Odds Ratio (OR) and 95% confidence interval (CI) of the blood pressure in mmHg.
Description of the risk factors for complications with the physiological parameters | 2011-2016
  We will study the increased risk of an event associated with a variable reported as the Odds Ratio (OR) and 95% confidence interval (CI) of the cardiac rate in bpm.
Description of the risk factors for complications with the physiological parameters | 2011-2016
  We will study the increased risk of an event associated with a variable reported as the Odds Ratio (OR) and 95% confidence interval (CI) of the respiratory rate in bpm.
Description of the risk factors for complications with the laboratory test | 2011-2016
  We will study the increased risk of an event associated with a variable reported as the Odds Ratio (OR) and 95% confidence interval (CI) of the bilirubin in mg/dL.
Description of the risk factors for complications with the laboratory test | 2011-2016
  We will study the increased risk of an event associated with a variable reported as the Odds Ratio (OR) and 95% confidence interval (CI) of the creatinine in mg/dL.
Description of the risk factors for complications with the laboratory test | 2011-2016
  We will study the increased risk of an event associated with a variable reported as the Odds Ratio (OR) and 95% confidence interval (CI) of the alkaline phosphatase in U/L.
Description of the risk factors for complications with the laboratory test | 2011-2016
  We will study the increased risk of an event associated with a variable reported as the Odds Ratio (OR) and 95% confidence interval (CI) of the gamma-glutamyl-transferase in U/L.
Description of the risk factors for complications with the laboratory test | 2011-2016
  We will study the increased risk of an event associated with a variable reported as the Odds Ratio (OR) and 95% confidence interval (CI) of the glutamyl oxaloacetic transaminase in U/L.
Description of the risk factors for complications with the laboratory test | 2011-2016
  We will study the increased risk of an event associated with a variable reported as the Odds Ratio (OR) and 95% confidence interval (CI) of the protrombine Time-INR.
Description of the risk factors for complications with the laboratory test | 2011-2016
  We will study the increased risk of an event associated with a variable reported as the Odds Ratio (OR) and 95% confidence interval (CI) of the lactate in gr/dL.
Description of the risk factors for complications with the laboratory test | 2011-2016
  We will study the increased risk of an event associated with a variable reported as the Odds Ratio (OR) and 95% confidence interval (CI) of the White Blood Cell count.
Description of the risk factors for complications with the laboratory test | 2011-2016
  We will study the increased risk of an event associated with a variable reported as the Odds Ratio (OR) and 95% confidence interval (CI) of the partial oxygen pressure in mmHg.
Description of the risk factors for complications with the laboratory test | 2011-2016
  We will study the increased risk of an event associated with a variable reported as the Odds Ratio (OR) and 95% confidence interval (CI) of the C-Reactive Protein in gr/dL.
Description of the risk factors for complications with the laboratory test | 2011-2016
  We will study the increased risk of an event associated with a variable reported as the Odds Ratio (OR) and 95% confidence interval (CI) of the platelets count.
Description of the risk factors for complications with the grade of severity of ACC following the TG18 | 2011-2016
  We will study the increased risk of an event associated with a variable reported as the Odds Ratio (OR) and 95% confidence interval (CI) of the following variables:
  * Grade I or Mild ACC
  * Grade II or Moderate ACC
  * Grade III or Severe ACC
Description of the risk factors for complications with the grade of severity of ACC following the Charlson Comorbidity Index | 2011-2016
  We will study the increased risk of an event associated with a variable reported as the Odds Ratio (OR) and 95% confidence interval (CI) of the following the charlson comorbidity index in two groups: above 6 and below 6.
Description of the risk factors for complications with the ASA Classification | 2011-2016
  We will study the increased risk of an event associated with a variable reported as the Odds Ratio (OR) and 95% confidence interval (CI) of the following the charlson comorbidity index in two groups:
  * Group I and II
  * Group III and IV

CONTACTS AND LOCATIONS:
Overall Officials: Ana María González-Castillo, M.D., Principal Investigator — Hospital del Mar

IPD SHARING:
Plan to Share IPD: Yes
all primary and secondary variables of anonymized individual data set will be provided
Time Frame: May 2021 to May 2022
Access Criteria: any researcher